CLINICAL TRIAL: NCT03685890
Title: A Phase Ib/II Randomized Double-blind Placebo Controlled Trial Evaluating the Effect of Nivolumab for Patients With In-transit Melanoma Metastases Treated With Isolated Limb Perfusion - the NivoILP Trial
Brief Title: Evaluating the Effect of Nivolumab for Patients With In-transit Metastases Treated With Isolated Limb Perfusion
Acronym: NivoILP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, Associate professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUGBG-KIR-2018-001
Record Dates: First submitted 2018-09-23; First posted 2018-09-26 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Melanoma; In-Transit Metastasis
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: The study is a randomized placebo controlled double blind trial. Patients will be randomized to ILP with nivolumab or ILP with placebo. Active follow-up for 3 years.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ILP + Nivolumab (Experimental): The day before planned ILP, the patient will receive one infusion of nivolumab 480mg
  Interventions: Drug: Nivolumab; Procedure: Isolated limb perfusion (ILP)
- ILP + Placebo (Placebo Comparator): The day before planned ILP, the patient will receive one infusion of placebo
  Interventions: Procedure: Isolated limb perfusion (ILP)

INTERVENTIONS:
Drug: Nivolumab — One infusion of nivolumab (Opdivo®) 480mg (flat dose) in NaCl (Natriumklorid Baxter Viaflo, 9 mg/ml) during 60 minutes
  Arms: ILP + Nivolumab
Procedure: Isolated limb perfusion (ILP) — Patients will be treated with ILP according to clinical routine at each separate site. The procedure is performed under general anaesthesia. The major artery and vein of the limb is catheterized, and a tourniquet is placed proximally on the limb. Continuous leakage monitoring is performed. The perfusate is heated to 40C and after ensuring steady state, melphalan (Alkeran®) at a dose of 13 mg/L (upper limb) or 10 mg/L (lower limb) is infused into the circulation during 20 minutes for a total perfusion time of 60 minutes. According to local routine tasonermin (Beromun®) will be added to the perfusate 30 minutes before the melphalan as a bolus dose of 1-4 mg.

SUMMARY:
To evaluate safety and the effect of isolated limb perfusion together with nivolumab as a way to increase efficacy and give further insights in early immunological mechanisms.

In the first phase Ib part, 20 patients will be enrolled and followed for a minimum of 3 months. An independent data safety monitoring board (DSMB) will continuously review safety and judge the seriousness of the events and also recommend the study to stop if necessary. If the DSMB do not find safety issues, the trial will continue as a phase II trial.

ELIGIBILITY:
Inclusion Criteria

1. Male or female aged above 18 years.
2. Signed and dated written informed consent before the start of specific protocol procedures.
3. Histologically or cytologically proven in-transit metastases of malignant melanoma with or without regional lymph node metastases (AJCC v8 stage N1c, N2c and N3c).
4. Measurable disease with at least 1 metastasis measuring at least 5mm
5. ECOG performance status of 0-2

Exclusion Criteria

1. 1. Life expectancy of less than 6 months
2. Inability to understand given information or undergo study procedures according to protocol.
3. Pregnant or breast-feeding. Women of childbearing potential must have a negative pregnancy test performed within 24 hours before the administration of study drug.
4. Patients must agree to follow instructions for method of contraception for 5 months (women) and 7 months (males) after treatment.
5. Active cardiac conditions, including unstable coronary syndromes (unstable or severe angina, recent myocardial infarction), significant arrhythmias and severe valvular disease that precludes general anaesthesia.
6. History or evidence of clinically significant pulmonary disease e.g., severe COPD that precludes general anesthesia.
7. Reduced renal function defined as S-Creatinine >=1.5xULN
8. Reduced hepatic function (defined as ASAT, ALAT, bilirubin >1.5 ULN and PK-INR >1.5) or a medical history of liver cirrhosis or portal hypertension.
9. Reduced blood leukocytes or platelets defined as a leucocyte count < 2.0x109/L and thrombocyte count <100x109/L.
10. Active, autoimmune disease. Subjects are permitted to enrolment if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
11. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
12. A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 30 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted.
13. Has an active infection requiring systemic therapy.
14. Has received a live vaccine within 30 days prior to the first dose of trial treatment and 3 months after treatment.
15. Concomitant therapy with any of the following: IL 2 or other non-study immunotherapy regimens; cytotoxic chemotherapy except melphalan (ILP); other investigational therapies within 30 days before trial treatment and 3 months after trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CR) | 3 months
  To evaluate if melphalan based isolated limb perfusion (ILP) synergizes with nivolumab in inducing complete responses (CR) at 3 months after treatment in melanoma patients with in-transit metastasis.

SECONDARY OUTCOMES:
Time to local progression (TTLP) | 36 months
  Evaluation of local progression-free survival (LPFS). LPFS is defined as the number of months from the date of ILP to the date of the first documented disease recurrence or progression in the treated area (defined as the area below the tourniquet used for ILP). LPFS will be determined based on clinical assessments according to RECIST version 1.1 criteria.
Distant metastases-free survival (DMFS) | 36 months
  Evaluation of DMFS, defined as the number of months from the date of ILP to the date of the first documented distant disease recurrence.
Progression-free survival (PFS) | 36 months
  Evaluation of PFS, defined as the number of months from the date of ILP to the date of the first documented disease recurrence or progression at any site.
Melanoma specific survival (MSS) | 36 months
  Evaluation of melanoma specific survival (MSS), MSS is calculated as the time from date of treatment to date of death due to any cause. Both median MSS and the per cent of patients alive at 36 months will be evaluated.
Overall survival (OS) | 36 months
  Evaluation of overall survival (OS), OS is calculated as the time from date of treatment to date of death due to any cause. Both median OS and the per cent of patients alive at 36 months will be evaluated.
Quality of life measured by FACT-M | 36 months
  Quality of life (QoL) by FACT-M. Change from baseline for all subscales as well as for the total scores.
Quality of life measured by EQ-5D | 36 months
  Quality of life (QoL) by EQ-5D measured as the change from baseline

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (3):
  - Netherlands Cancer Institute, Amsterdam
  - Erasmus MC Cancer Institute, Groningen
  - Erasmus MC Cancer Institute, Rotterdam
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Holmberg CJ, Zijlker LP, Katsarelias D, Huibers AE, Wouters MWJM, Schrage Y, Reijers SJM, van Thienen JV, Grunhagen DJ, Martner A, Nilsson JA, van Akkooi ACJ, Ny L, van Houdt WJ, Olofsson Bagge R. The effect of a single dose of nivolumab prior to isolated limb perfusion for patients with in-transit melanoma metastases: An interim analysis of a phase Ib/II randomized double-blind placebo-controlled trial (NivoILP trial). Eur J Surg Oncol. 2024 Jun;50(6):108265. doi: 10.1016/j.ejso.2024.108265. Epub 2024 Mar 12. PMID 38493679
- [Derived] Constantinescu A, Olofsson Bagge R, Huibers A. Immunological phenotype as a predictor for response after isolated limb perfusion for patients with melanoma in-transit metastasis. Eur J Surg Oncol. 2026 Jan 23;52(3):111424. doi: 10.1016/j.ejso.2026.111424. Online ahead of print. PMID 41616426
- [Derived] Tulokas SKA, Kohtamaki LM, Makela SP, Juteau S, Alback A, Vikatmaa PJ, Mattila KE, Skytta TK, Koivunen JP, Tyynela-Korhonen K, Hernberg MM. Isolated limb perfusion with melphalan as treatment for regionally advanced melanoma of the limbs: results of 60 patients treated in Finland during 2007-2018. Melanoma Res. 2021 Oct 1;31(5):456-463. doi: 10.1097/CMR.0000000000000755. PMID 34132224